CLINICAL TRIAL: NCT04227366
Title: An International, Multicenter, Randomized, Double-blind, Placebo-controlled Clinical Study of the Efficacy and Safety of BCD-089 (JSC BIOCAD, Russia) in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis
Brief Title: Study of the Efficacy and Safety of BCD-089 in Combination With Methotrexate in Patients With Active Rheumatoid Arthritis
Acronym: SOLAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCD-089-3
Record Dates: First submitted 2019-12-25; First posted 2020-01-13 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2020-11

CONDITIONS: Rheumatoid Arthritis
Keywords: anti-IL-6R; IL-6 receptor inhibitors
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — levilimab; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): BCD-089
  Interventions: Biological: BCD-089; Drug: Methotrexat
- Group 2 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo; Drug: Methotrexat

INTERVENTIONS:
Biological: BCD-089 — BCD-089 162 mg SC
  Arms: Group 1
Biological: Placebo — Placebo
  Other Names: Placebo (for BCD-089)
  Arms: Group 2
Drug: Methotrexat — 15 to 25 mg/week

SUMMARY:
BCD-089 is the original therapeutic monoclonal antibody binding the alpha subunit of the IL-6 receptor.

The aim of the study is to demonstrate the efficacy and safety of BCD-089 in combination with methotrexate in patients with active rheumatoid arthritis resistant to monotherapy with methotrexate.

DETAILED DESCRIPTION:
BCD-089-3/SOLAR is the international, multicenter, double blind, placebo-controlled phase III clinical study.

The main period of the study (Weeks 0-24) is blinded; study subjects will receive BCD-089/placebo.

At Week 24 the study will become open-label and all patients will receive BCD-089 once a week for 4 weeks. At week 28 patients who achieved the RA remission at week 24 will be switched to BCD-089 Q2W dosing regimen and will receive it through Week 51. Patients who failed to achieve remission at week 24 will receive BCD-089 once a week through Week 51.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form (ICF).
2. Men and women aged 18 years or older on the day of signing the ICF.
3. Verified rheumatoid arthritis according to the ACR 2010 criteria diagnosed at least 24 weeks before signing the ICF .
4. Use of methotrexate for the last 12 weeks before signing the ICF.
5. Use of a stable dose of methotrexate for the last 4 weeks before signing the ICF (the dose of methotrexate should be 15 to 25 mg per week). Methotrexate can be used at a dose of 10 mg in the case of intolerability/toxicity of higher doses.
6. Inefficacy of methotrexate used for the last 12 weeks before signing the ICF (in the opinion of the Investigator).
7. Active rheumatoid arthritis at randomization in the study.
8. The ability of the patient (in the Investigator's opinion) to follow the Protocol procedures.
9. Patients and their sexual partners of childbearing potential agree to use reliable contraceptive methods starting from signing the ICF, during the study and for 8 weeks from the last injection of the investigational product. This requirement does not apply to patients and their partners who underwent surgical sterilization and to women who are post-menopausal for at least 2 years. Reliable contraceptive methods include one barrier method in combination with one of the following: spermicides, intrauterine device/oral contraceptives.

Exclusion Criteria:

1. Previous exposure to tocilizumab or other anti-IL6 or anti-IL-6R monoclonal antibodies.
2. Previous exposure to JAK inhibitors.
3. Previous exposure to rituximab or other B-cell depleting/suppressing agents.
4. Felty's syndrome (regardless of clinical form).
5. Patient's functional status: class IV according to the ACR 1991 classification.
6. Known allergy to or intolerance of any ingredients of BCD-089 or placebo.
7. Use of any of the following concomitant therapies:

   * Oral prednisolone or its equivalent in a dose more than 10 mg/day;
   * Need in oral prednisolone (or its equivalent) ≤ 10 mg if its dose was not stable during the last 4 weeks before signing the ICF (patients who used topical glucocorticoids are allowed to participate in the study);
   * Need in NSAIDs if the dose was not stable during the last 4 weeks before signing the ICF (patients who have occasionally used NSAIDs for fever or allergy syndrome associated with an intercurrent disease can be included in the study);
   * Use of alkylating agents any time within 12 months before signing the ICF.
   * Intra-articular use of corticosteroids within 4 weeks before signing the ICF.
   * Vaccination with live or attenuated vaccines any time within 8 weeks before signing the ICF.
   * Use of leflunomide within 8 weeks before signing the ICF.
   * Use of TNFα inhibitors or T-cell costimulation blockers within 8 weeks before signing the ICF.
8. Any of the following laboratory values at screening:

   * Hemoglobin level < 80 g/L;
   * Leukocyte count < 3.0 × 109/L;
   * Platelet count < 100 × 109/L;
   * Neutrophil count < 2 × 109/L;
   * AST and ALT ≥ 1.5×ULN (based on the reference limits used by the laboratory);
   * Serum creatinine ≥ 1.7 × ULN (based on the reference limits used by the laboratory).
9. Positive pregnancy urine test in female subjects at screening (no test is required in women who are post-menopausal for at least 2 years and in surgically sterile women).
10. Current diagnosis or a history of a severe immunodeficiency of any other origin.
11. Diagnosed HIV, hepatitis B, hepatitis C, or syphilis ;
12. Tuberculosis now or in the past.
13. Latent TB forms (positive Diaskintest®, QuantiFERON®-TB Gold or T-SPOT.TB test with no radiographic signs of pulmonary TB).
14. Herpes zoster infection now or in the past .
15. Documented chickenpox within 30 days before signing the ICF.
16. Definite diagnosis of any other chronic infection (e.g. sepsis, invasive mycoses, histoplasmosis, etc.) that, in the Investigator's opinion, can increase the risk of infectious complications.
17. Any acute infection or aggravation of a chronic infection within 30 days before signing the ICF if this condition may, in the Investigator's opinion, increase the risk of infectious complications.
18. Severe infections (including those that required hospitalization or parenteral antibacterial/antimycotic/antiprotozoal treatment) within 6 months before signing the ICF.
19. Systemic antibacterial/antimycotic/antiprotozoal treatments used within 8 weeks before the signing the ICF.
20. More than 4 episodes of respiratory infections within 6 months before signing the ICF.
21. A major surgery within 30 days before signing the ICF or a major surgery scheduled at any time during the study.
22. History of epileptic attacks or seizures.
23. History of severe depression, suicidal thoughts or suicide attempts .
24. Diverticulosis and/or diverticulitis .
25. Alcohol, drug or psychoactive substance dependence or medication abuse now or in the past, signs of alcohol/drug dependence.
26. Other documented medical conditions that can increase a risk of adverse events during the study treatment, affect the assessment of the main disease severity, mask, aggravate, affect symptoms of the main disease, or result in the same clinical and laboratory instrumental symptoms as those of rheumatoid arthritis:

    * Diabetes mellitus with inadequate glycemic control ;
    * Severe treatment-resistant hypertension ;
    * Current or a history of inflammatory joint diseases other than rheumatoid arthritis (including ankylosing spondylitis, gout, psoriatic arthritis, Lyme disease etc. ) or other systemic autoimmune diseases (including systemic lupus erythematosus, Crohn's disease, non-specific ulcerative colitis, systemic scleroderma, inflammatory myopathy, mixed connective tissue disease, overlap syndrome, fibromyalgia etc.);
    * Malignant neoplasms except for cured basal-cell carcinoma and cancer of the cervix in situ (complete remission ≥ 5 years); cured basal-cell carcinoma of the skin (complete remission ≥ 5 years); cured ductal breast cancer (complete remission ≥ 5 years);
    * Decompensated liver or kidney diseases;
    * Unstable angina;
    * Chronic heart failure of NYHA class III-IV;
    * Myocardial infarction within 1 year before signing the ICF;
    * History of organ transplantation;
    * History of angioedema;
    * Respiratory system disorders with decompensated respiratory insufficiency;
    * Definite diagnosis of multiple sclerosis, Devic's disease, or Guillain-Barre syndrome;
    * Nervous system disorders with motor and/or sensitivity abnormalities.
27. Pregnancy , planned pregnancy less than 8 weeks after the last injection of the investigational product; lactation.
28. Current participation in other clinical studies; previous participation in other clinical studies within 3 calendar months before signing the ICF (except for screenouts); previous participation in this study (except for screenouts).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2019-11-19 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
ACR 20 response | Week 12
  The proportion of ACR 20 responders
Low disease activity | Week 24
  The proportion of patients with low disease activity according to DAS28-CRP(4) (< 3,2)

SECONDARY OUTCOMES:
Need for rescue therapy | Week 12.
  The proportion of patients who required rescue therapy
RA remission | Weeks 4, 8, 12, 16, 24.
  The proportion of patients who achieved RA remission according to DAS28-CRP(4) (< 2.6)
RA remission | Weeks 4, 8, 12, 16, 24.
  The proportion of patients who achieved RA remission according to CDAI (≤ 2.8)
RA remission | Weeks 4, 8, 12, 16, 24.
  The proportion of patients who achieved RA remission according to SDAI (≤ 3.3)
Remission according to the ACR/EULAR 2011 criteria | Weeks 4, 8, 12, 16, 24
  The proportion of patients who achieved remission
ACR20 response | Weeks 4, 8, 16, 24
  The proportion of ACR20 responders
ACR50 response | Weeks 4, 8, 12, 16, 24
  The proportion of ACR50 responders
ACR70 response | Weeks 4, 8, 12, 16, 24
  The proportion of ACR70 responders
Low RA activity according to DAS28-ESR(4) | Weeks 4, 8, 12, 16, 24
  The proportion of patients who achieved low RA activity according to DAS28-ESR(4) (< 3.2)
Low RA activity according to CDAI | Weeks 4, 8, 12, 16, 24.
  the proportion of patients who achieved low RA activity according to CDAI (≤ 10)
Low RA activity according to SDAI | Weeks 4, 8, 12, 16, 24.
  The proportion of patients who achieved low RA activity according to SDAI (≤ 11)
Change in the DAS28-CRP(4) | Weeks 4, 8, 12, 16, 24.
  The change from baseline in the DAS28-CRP(4)
Change in the CDAI | Weeks 4, 8, 12, 16, 24.
  The change from baseline in the CDAI
Change in the SDAI | Weeks 4, 8, 12, 16, 24.
  The change from baseline in the SDAI
Moderate/good response according to the EULAR criteria | Weeks 4, 8, 12, 16, 24
  The proportion of patients with moderate/good response according to the EULAR criteria
Change in concentration of C-reactive protein | Weeks 4, 8, 12, 16, 24.
  The change from baseline in the concentration of C-reactive protein in serum
Change in the ESR | Weeks 4, 8, 12, 16, 24
  The change from baseline in the erythrocyte sedimentation rate (ESR)
Change in the quality of life measured with SF-36 | Weeks 12, 24
  The change from baseline in the patient's quality of life measured with the SF-36 score
Change in the quality of life measured with the EQ-5D-3L | Weeks 12, 24
  The change from baseline in the patient's quality of life measured with the EQ-5D-3L
Change in the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) score | Weeks 12, 24
  The change in the FACIT-F score. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued) (Webster et al., 2003)
Change in functional activity | Weeks 12, 24
  The change in functional activity according to the HAQ-DI (Health Assessment Questionnaire without Didability Index) score. The value of the HAQ-DI index can be interpreted in terms of three categories:
  from 0 to 1: mild difficulties to moderate disability, from 1 to 2: disability moderate to severe, from 2 to 3: severe to very severe disability.
X-ray assessment | Week 24
  The change in mTSS score according to Sharp/van der Heijde (SvH) scoring method

CONTACTS AND LOCATIONS:
Overall Officials: Yulia Linkova, MD, PhD, Study Chair — JSC BIOCAD
Locations (1):
- Research Institute of Rheumotology, Moscow, Russia

REFERENCES:
- [Background] Mazurov V.I., Korolev M.A., Prystrom A.M., Kunder E.V., Soroka N.F., Kastanayan A.A., Povarova T.V., Plaksina T.V., Antipova O.V., Kretchikova D.G., Smakotina S.A., Tciupa O.A., Puntus E.V., Raskina T.A., Shilova L.N., Kropotina T.V., Nesmeyanova O.B., Popova T.A., Vinogradova I.B., Linkova Yu.N., Dokukina E.A., Plotnikova A.V., Pukhtinskaia P.S., Zinkina-Orikhan A.V., Eremeeva A.V., Lutckii A.A. Effectiveness and safety of levilimab in combination with methotrexate in treatment of patients with active rheumatoid arthritis resistant to methotrexate monotherapy (double-blinded randomized placebo controlled phase III clinical study SOLAR). Modern Rheumatology Journal. 2021;15(4):13-23. https://doi.org/10.14412/1996-7012-2021-4-13-23
- See also: Related Info — https://mrj.ima-press.net/mrj/article/view/1164/1169